CLINICAL TRIAL: NCT05597397
Title: Effect of Repeated Low-Level Red-Light Therapy on Retinal Function and Structure Among Myopic Teenagers
Brief Title: Effect of Repeated Low-Level Red-Light Therapy on Retinal Function and Structure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RLS-SEPTC-2022
Record Dates: First submitted 2022-09-20; First posted 2022-10-28 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Myopia; Refractive Errors; Eye Diseases; Retina; Change
MeSH Terms: conditions — Myopia; Refractive Errors; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repeated Low-Level Red-Light Therapy (RLRL) (Experimental): Single vision spectacles (SVS) & RLRL.
  Interventions: Device: RLRL

INTERVENTIONS:
Device: RLRL — In addition to SVS with power for correcting distance refraction, RLRL will be performed twice per school day with an interval of at least 4 hours, each treatment last 3 minutes.

SUMMARY:
The purpose of this clinical trial is to evaluate the effect of repeated low-level red-light (RLRL) therapy on the retinal function and structure among myopic teenagers.

DETAILED DESCRIPTION:
Myopia constitutes a major threat to personal health globally for its increased prevalence. Moreover, its dose-related association with irreversible blindness complications such as myopic macular degeneration has been demonstrated. It is crucial to look for effective ways to control myopia in children to reduce risk of myopic pathologies in later life. Repeated low-level red-light (RLRL) therapy is an innovative and non-invasive therapeutic treatment for a variety of eye diseases. A previous randomized clinical trial suggested that RLRL could effectively controlled myopia progression without clinically observable side effects.

The purpose of this study is to evaluate the effect of RLRL on the retinal function and structure among myopic teenagers aged 15-16 years. The RLRL therapy will be carried out at school under supervision of the parents according to a standard protocol for the first month and then will be discontinued for 1 month. Detailed functional and structural examinations, including full field electroretinogram, multifocal electroretinogram, microperimetry, visual acuity, intraocular pressure, optical coherence tomography, optical coherence tomography angiography, cycloplegic spherical equivalent refraction, and biological parameters will be evaluated at 1 month, 2 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 15-16 years at enrolment.
2. Myopia: cycloplegic spherical equivalent refractions (SERs) range from -1.00 to -5.00 diopters (D) and astigmatism less than -2.5 D in either eye.
3. Best corrected visual acuity equal to or better than 0.8 in either eye.
4. Normal fundus, or tessellated fundus.
5. Provision of consent and able to participate in all required activities of the study.

Exclusion Criteria:

1. Secondary myopia, such as a history of retinopathy of prematurity or neonatal problems, or syndromic myopia with a known genetic disease or connective tissue disorders, such as Stickler or Marfan syndrome.
2. Strabismus and binocular vision abnormalities in either eye.
3. Refractive media opacity: corneal opacities, cataract, or implanted intraocular lens, etc.
4. Ocular abnormalities that affect retinal function: macular degeneration, diabetic retinopathy, retinal detachment, glaucoma, or ocular hypertension, endophthalmitis, uveitis, optic neuropathy, etc.
5. Previous history of refractive surgery, intraocular surgery, laser therapy, and intravitreal injection, etc.
6. Systemic abnormalities: diabetes, hypertension, etc.
7. Drugs therapies with toxicity effect on the retina: hydroxychloroquine, etc.
8. Prior treatment of myopia control in the past three months, drugs, orthokeratology, progressive addition lenses, bifocal lens, etc.
9. Other contraindications, including but not limited to ocular or other systemic abnormalities, that the physician may consider inappropriate for enrolment.

Ages: 15 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Changes in the amplitudes of waves. | 1 and 2 months
  Changes in the amplitudes are characterized as the difference between each follow-up visit and corresponding baseline values which are measured by electroretinogram.
Changes in the latency of waves. | 1 and 2 months
  Changes in the latency of waves are characterized as the difference between each follow-up visit and corresponding baseline values which are measured by electroretinogram.

SECONDARY OUTCOMES:
Changes in retinal sensitivity | 1 and 2 months
  Changes in retinal sensitivity are characterized as the difference between each follow-up visit and corresponding baseline values which are measured by microperimetry.
Changes in fixation stability | 1 and 2 months
  Changes in fixation stability are characterized as the difference between each follow-up visit and corresponding baseline values which are measured by microperimetry.
Changes in macular integrity | 1 and 2 months
  Changes in macular integrity are characterized as the difference between each follow-up visit and corresponding baseline values which are measured by microperimetry.
Changes in macular vessel density | 1 and 2 months
  Changes in macular vessel density are characterized as the difference between each follow-up visit and corresponding baseline values which are measured by optical coherence tomography angiography.
Changes in macular perfusion density | 1 and 2 months
  Changes in macular perfusion density are characterized as the difference between each follow-up visit and corresponding baseline values which are measured by optical coherence tomography angiography.
Changes in chorocapillaris flow defict percentage | 1 and 2 months
  Changes in choroidal vascularity index are characterized as the difference between each follow-up visit and corresponding baseline values which are measured by optical coherence tomography angiography.
Changes in choroidal vascularity index | 1 and 2 months
  Changes in choroidal vascularity index are characterized as the difference between each follow-up visit and corresponding baseline values which are measured by optical coherence tomography.
Changes in best corrected visual acuity | 1 and 2 months
  Best corrected visual acuity changes are characterized as the difference between each follow up visit and baseline values. An Early Treatment Diabetic Retinopathy Study chart with standard illumination at a distance of 4 meters is used to measure best corrected visual acuity.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as open data after proper anonymization.